CLINICAL TRIAL: NCT01817218
Title: Feasibility and Safety and Evaluation of the Potential Efficacy of Autologous Platelet-rich Plasma in the Treatment of Vascular Venous Ulcers Compared to Moist Wound Care in a Primary Care Setting
Brief Title: Feasibility and Safety and Evaluation of the Potential Efficacy of Autologous Platelet-rich Plasma in the Treatment of Vascular Venous Ulcers
Acronym: PRP-2012
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Kepa M. San Sebastián Moreno, Dr., Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-002247-20
Record Dates: First submitted 2013-02-27; First posted 2013-03-25 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Ulcer
Keywords: PRP; chronic vascular ulcer; primary care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRP (Platelet Rich Plasma) (Experimental): PRP treatment of vascular ulcers one a week PRP: a volume of 9-30 ml of blood will be collected from the patient (depending of the size of their ulcer) in sterile 4.5-ml tubes containing 3.8% sodium citrate, which will bind to the calcium ions, preventing clot formation we will add 50 μl of CaCl2 per ml liquid plasma. The extraction of the PRP fraction by sticking with a syringe and the adding of CaCl2 should be performed under sterile conditions.
  Interventions: Drug: Platelet Rich Plasma
- Osakidetza protocol (Active Comparator): Patients in the control group will be treated following the recommendations of the Ezkerraldea-Enkarterri Health Region, that is, using a moist healing environment (as described in "Uso racional de los productos de cura en ambiente húmedo. Plan de formación continuada de Osakidetza", 2011).
  The type of material used to treat and dress the wound will be chosen after the assessment of the wound and surrounding skin, type and quantity of exudate and whether there are signs of infection. Wound care will be carried out every 48-72 hours, as is the current usual practice.
  Interventions: Device: Osakidetza protocol

INTERVENTIONS:
Drug: Platelet Rich Plasma
  Arms: PRP (Platelet Rich Plasma)
Device: Osakidetza protocol — Patients in the control group will be treated following the recommendations of the Ezkerraldea-Enkarterri Health Region, that is, using a moist healing environment (as described in "Uso racional de los productos de cura en ambiente húmedo. Plan de formación continuada de Osakidetza", 2011).
  The type of material used to treat and dress the wound will be chosen after the assessment of the wound and surrounding skin, type and quantity of exudate and whether there are signs of infection. Wound care will be carried out every 48-72 hours, as is the current usual practice.
  Other Names: "Antimicrobial debridin"; "hydrocolloids"; "alginates and hydrofibres"; "polyurethane foams"; "barrier products"
  Arms: Osakidetza protocol

SUMMARY:
INTRODUCTION: Vascular ulcers are an important pathology in the daily medical practice in all the assistance levels, and they have big repercussion referring to individual, social and labour levels, supposing a big consumption of human and material resources.The cure with autologous platelet rich plasma (autologous PRP) has demonstrated in different studies a decrease in the cicatrization time comparing to conventional methods in hospital levels, which becomes interesting contrasting its efficacy in primary care.

AIM:Evaluate the practicability, security and potential of the autologous PRP in the treatment of vascular ulcers, comparing to the conventional treatment ( cure with humid environment), in primary care patients with chronic venous insufficiency in C-6 degree (CEAP classification).

DESIGN:A pilot study will be executed, which will consist in a randomized clinical test, multicentred, in parallel groups and opened. 40 patients suffering of venous vascular ulcers will be studied, who will be between the age of 40-80 years old, and who will be attached to five health centers. Variables for the identification, following, result and patient profile have been defined. Emphasize the variables of "ulcer area decreasing", "CIVIQ index", "% one cure per week" .

ELIGIBILITY:
Inclusion Criteria:

* Patients resident in Barakaldo, who are seen in treatment rooms at the Zaballa outpatient clinic or one of the following health centres: Zaballa, La Paz, Urban, or San Vicente, in the Ezkerraldea-Enkarterri Health Region of the Basque Health Service - Osakidetza.
* Men or women of 40 to100 years of age
* Patients with stage C6 chronic venous insufficiency according to the CEAP classification
* Patients with vascular ulcers which have not responded to conventional treatment in 2 to 6 months
* Patients who present an analytical before entering the study with a normal range of number of platelets, red blood cells and hematocrit
* An ulcer of 3-5 cm in diameter
* An ABI of greater than or equal to 0.8 or less than or equal to 1.5.
* Independent patients or with sufficient family support
* Patients have given written informed consent

Exclusion Criteria:

* Patients with chronic treatment with immunosuppressive or retroviral drugs
* Coagulopathies
* Patients with chronic infectious diseases
* Patients under radiotherapy or chemotherapy
* Patients with a history of neoplasia
* Patients with more than two active ulcers
* Pregnant women
* Patients with active cellulitis or fever
* An ABI of less than 0.8 or more than 1.5.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change of ULCER AREA | Change from baseline at 9 weeks
  Change from baseline at 9 weeks of the surface area of the ulcer, in cm3, measured using ImageJ software from the weekly the photographs of the wound
Change of the percentage OF PATIENTS WITH A ONLY ONE TREATMENT FOR WEEK | Change from baseline at 9 weeks
  Change of the percentage OF PATIENTS WITH A ONLY ONE TREATMENT FOR WEEK
REDUCTION IN ULCER SIZE | Change from baseline at 9 weeks
  Difference in the area of the wound between week 9 and the first treatment session.
Change of the CIVIQ SCORE | Change from baseline to 9th week
  change of the scale assessing quality of life of patients with chronic venous insufficiency, considering four dimensions (physical, psychological, social and pain) with a score ranging from 20 to 100, where 20 corresponds to the poorest quality of life and 100 to the best.

CONTACTS AND LOCATIONS:
Overall Officials: Kepa Mirena San Sebastian Moreno, Doctor, Principal Investigator — Osakidetza
Locations (1):
- Comarca Enkarterri Ezkerraldea, Portugalete, Bizakaia, Spain